CLINICAL TRIAL: NCT04233567
Title: A Phase II Study of Oral Infigratinib in Adult Patients With Advanced or Metastatic Solid Tumors With FGFR1-3 Gene Fusions or Other FGFR Genetic Alterations
Brief Title: Infigratinib for the Treatment of Advanced or Metastatic Solid Tumors in Patients With FGFR Gene Mutations
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sameek Roychowdhury (Other)
Responsible Party: Sponsor-Investigator, Sameek Roychowdhury, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19041; NCI-2019-06869 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Advanced Malignant Solid Neoplasm; Cholangiocarcinoma; Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasm Metastasis | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (infigratinib) (Experimental): Patients receive infigratinib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Infigratinib

INTERVENTIONS:
Drug: Infigratinib — Given PO
  Other Names: 3-(2,6-Dichloro-3,5-dimethoxyphenyl)-1-(6-((4-(4-ethylpiperazin-1-yl)phenyl)amino)pyrimidin-4-yl)-1-methylurea; BGJ-398; BGJ398

SUMMARY:
This phase II trial studies how well infigratinib works in treating solid tumors that have spread to other places in the body (advanced or metastatic) in patients with FGFR gene mutations such as FGFR1-3 gene fusions or other FGFR genetic alterations. Mutations are any changes in the genetic material (DNA) of a cell. FGFR proteins are involved in cell division, cell maturation, formation of new blood vessels, wound healing, and bone growth, development, and maintenance. FGFR mutations can cause the FGFR protein to become over-active in diseases such as cancer. Infigratinib may stop the growth of tumor cells by blocking FGFR proteins in these tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of single agent infigratinib in patients with advanced or metastatic solid tumors of any histologic classification with FGFR1-3 gene fusions/translocations or other FGFR genetic alterations (with and without prior therapy with different FGFR inhibitor).

II. To understand response rate and potential for infigratinib to benefit patients who have FGFR alterations including point mutations, insertions/deletions and amplifications in different solid tumor types.

SECONDARY OBJECTIVES:

I. To further evaluate the efficacy of single agent infigratinib. II. To characterize the safety and tolerability of single agent infigratinib. II. To evaluate benefit of infigratinib in patients who have received one prior FGFR inhibitor.

EXPLORATORY OBJECTIVES:

I. To detect biomarkers of resistance to infigratinib treatment through tumor sequencing.

II. To develop a circulating tumor deoxyribonucleic acid (DNA) (ctDNA) or liquid biopsy assay optimized for monitoring response to infigratinib and detecting emerging resistance mutations to infigratinib.

OUTLINE:

Patients receive infigratinib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients who complete study treatment for any reason other than disease progression are followed for 30 days, every 8 weeks until disease progression, and then every 4 months for 1 year. All other patients are followed for 30 days, and then every 4 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced or metastatic solid tumors of any histologic classification at the time of diagnosis
* Written documentation of local or central Clinical Laboratory Improvement Act (CLIA)-certified laboratory determination of FGFR gene fusions/translocations or activating mutations
* The study is open to solid tumors in the following cohorts:

  * Cohort 1: Solid tumor patients with FGFR1-3 fusion/translocation (n=10) who have progressed on or are intolerant to standard of care (SOC) therapies and received treatment with a different FGFR inhibitor. Cholangiocarcinoma patients are permitted in this cohort
  * Cohort 2: Solid tumor patients with FGFR1-3 fusion/translocation (n, up to 30) who have progressed on or are intolerant to SOC therapies. Prior therapy with a different FGFR inhibitor is not permitted. Cholangiocarcinoma patients are excluded from this cohort (there are multiple competing studies and opportunities for patients to get treatment in other trials)
  * Cohort 3: Solid tumor patients with genetic alterations such as point mutations, insertions/deletions, or amplifications in any FGFR gene family member (n=10). Prior therapy with a different FGFR inhibitor is not permitted. Cholangiocarcinoma patients are permitted in this cohort
* Evidence of measurable or evaluable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Patients must have received at least one prior SOC regimen for advanced/metastatic cancer. Patient should have had evidence of progressive disease following their prior regimen, or if prior treatment was discontinued due to toxicity must have continued evidence of measurable or evaluable disease. Patients who have received prior treatment with an alternate FGFR inhibitor are still eligible for the study
* Patients with primary central nervous system (CNS) cancer or CNS metastases are excluded (because it is unclear how much CNS penetration the drug has). However, asymptomatic patients with history of successfully treated CNS metastases with surgery or radiation and follow up imaging showing stability, can be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (patients with ECOG performance status of 2 may be considered on a case-by-case basis after discussion with QED Therapeutics)
* Able to read and/or understand the details of the study and provide written evidence of informed consent as approved by Institutional Review Board (IRB)/Ethics Committee (EC)
* Recovery from adverse events of previous systemic anti-cancer therapies to baseline or grade 1, except for:

  * Alopecia
  * Stable neuropathy of =< grade 2 due to prior cancer therapy
* Able to swallow and retain oral medication
* Willing and able to comply with scheduled visits, treatment plan and laboratory tests

Exclusion Criteria:

* Patients who have therapies available that are known to confer a clinical benefit will be excluded from the study
* Neurological symptoms related to underlying disease requiring increasing doses of corticosteroids. Note: Steroid use for management of CNS tumors is allowed but must be at a stable dose for at least 2 weeks preceding study entry
* History of another primary malignancy except adequately treated in situ carcinoma of the cervix or non-melanoma carcinoma of the skin or any other curatively treated malignancy that is not expected to require treatment for recurrence during the course of the study or affect survival
* Any other medical condition that would, in the investigator's judgment, prevent the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures
* Current evidence of corneal or retinal disorder/keratopathy including, but not limited to, bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, confirmed by ophthalmologic examination
* History and/or current evidence of extensive tissue calcification including, but not limited to, the soft tissue, kidneys, intestine, myocardium and lung with the exception of calcified lymph nodes, minor pulmonary parenchymal calcifications, and asymptomatic coronary calcification
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral infigratinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection)
* Current evidence of endocrine alterations of calcium/phosphate homeostasis, e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, tumoral calcinosis etc
* Treatment with any of the following anti-cancer therapies prior to the first dose of infigratinib within the stated timeframes:

  * Cyclical chemotherapy (intravenous) within a period of time that is shorter than the cycle length used for that treatment (e.g., 6 weeks for nitrosourea, mitomycin-C)
  * Biological therapy (e.g., antibodies - including bevacizumab) within a period of time that is =< 5 half-life (t1/2) or =< 4 weeks, whichever is shorter, prior to starting study drug
  * Continuous or intermittent small molecule therapeutics within a period of time that is =< 5 t1/2 or =< 4 weeks (whichever is shorter) prior to starting study drug
  * Any other investigational agents within a period of time that is =< 5 t1/2 or less than the cycle length used for that treatment or =< 4 weeks (whichever is shortest) prior to starting study drug
  * Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug
* Patients who are currently receiving treatment with agents that are known strong inducers or inhibitors of CYP3A4 and medications which increase serum phosphorus and/or calcium concentration are excluded. Patients are not permitted to receive enzyme-inducing anti-epileptic drugs
* Consumption of grapefruit, grapefruit juice, grapefruit hybrids, pomegranates, star fruits, pomelos, Seville oranges or products within 7 days prior to first dose
* Use of medications that are known to prolong the QT interval and/or are associated with a risk of Torsades de Pointes (TdP) 7 days prior to first dose
* Use of amiodarone within 90 days prior to first dose
* Current use of therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulants. Heparin and/or low molecular weight heparins are allowed
* Absolute neutrophil count (ANC) =< 1,000/mm^3 (1.0 x 10^9/L)
* Platelets =< 75,000/mm^3 (75 x 10^9/L)
* Hemoglobin =< 9.0 g/dL
* Total bilirubin >= 1.5 x upper limit of normal (ULN) unless associated with patient's primary cancer and/or metastases and with principal investigator's approval
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >= 3 x ULN unless associated with patient's primary cancer and/or metastases and with principal investigator's approval
* Alkaline phosphatase >= 2.5 x ULN unless associated with patient's primary cancer and/or metastases and with principal investigator's approval
* Calculated or measured creatinine clearance of < 40 mL/min
* Calcium-phosphate homeostasis:

  * Inorganic phosphorus outside of institutional normal limits
  * Total serum calcium (can be corrected) outside of institutional normal limits
* Clinically significant cardiac disease including any of the following:

  * Congestive heart failure requiring treatment (New York Heart Association [NYHA] grade >= 2), left ventricular ejection fraction (LVEF) < 50% as determined by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO), or uncontrolled hypertension (refer to World Health Organization [WHO] and International Society for Hypertension [ISH] guidelines)
  * History or presence of clinically significant ventricular arrhythmias, atrial fibrillation, resting bradycardia, or conduction abnormality
  * Unstable angina pectoris or acute myocardial infarction =< 3 months prior to starting study drug
  * Corrected QT using Fridericia's formula (QTcF) > 470 msec (males and females)
  * History of congenital long QT syndrome
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months following the discontinuation of study treatment. Highly effective contraception methods include:

  * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient
  * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine systems (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
  * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential
* Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of the study drug and should not father a child in this period. A condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2025-12-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sameek Roychowdhury, M.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Infigratinib)
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Infigratinib)
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Assessed by investigator as per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. The estimated ORR will be presented along with the corresponding 90% confidence interval for each cohort, based on a binomial distribution. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions: Complete Response (CR), Disappearance of all non-nodal target lesions; Partial Response (PR), at least a 30% decrease in the sum of diameter of all target lesions; Overall Response (OR) = CR + PR
Time Frame: 6 cycles of treatment (each cycle is 28 days) or upon treatment discontinuation
Population: Only 15 patients were evaluable for this outcome measure
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Infigratinib)
Number analyzed (Participants) | 15
percentage of participants | 13.3 [3.6 to 36.1]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Assessed by investigator as per RECIST v1.1. Kaplan-Meier analysis of PFS will be conducted for each cohort.
Time Frame: From start of treatment to the date of the event defined as the first documented progression or death due to any cause, assessed up to 1 year post-treatment, up to 5 years
Population: Only 15 patients were evaluable for this outcome measure
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Infigratinib)
Number analyzed (Participants) | 15
months | 3.73 [1.87 to 7.1]

3. Secondary Outcome: Disease Control Rate
Description: Assessed by investigator as per RECIST v1.1.
Time Frame: Up to 1 year post-treatment, up to 5 years
Population: Only 15 patients were evaluable for this outcome measure
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Infigratinib)
Number analyzed (Participants) | 15
percentage of participants | 73.3 [50 to 87.8]

4. Secondary Outcome: Overall Survival (OS)
Description: Assessed by investigator as per RECIST v1.1. Will be analyzed using the Kaplan Meier method. Survival rate at 4, 6, 8, 12, 18 and 24 months and median OS will be estimated along with 95% confidence intervals from the Kaplan Meier distribution.
Time Frame: From the date of start of treatment to the date of death due to any cause, will be assessed at 4, 6, 8,12 and 24 months
Population: Only 15 patients were evaluable for this outcome measure
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Infigratinib)
Number analyzed (Participants) | 15
months | 9.37 [3.97 to 12.5]

5. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: Will be tabulated and presented. All AEs occurring during the study will be included in by-patient data listings and tabulated by organ class and preferred term. Adverse events will be summarized overall, by relationship and by severity. Events leading to death, serious (S)AE, and events resulting in treatment discontinuation will be tabulated. Individual patient laboratory parameter values and summary statistics over time will be prepared using descriptive statistics. Severity of select clinical laboratory measures will be determined using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5 criteria .
Time Frame: Up to 30 days post-treatment, up to 5 years
Measure: Number; unit: events
Arm/Group | Treatment (Infigratinib)
Number analyzed (Participants) | 17
events
  Abdominal Cramping | 1
  Abdominal Pain | 18
  Alanine Aminotransferase Increased | 1
  Alkaline Phosphatase Increased | 3
  Allergic Reaction | 1
  Allergic Rhinitis | 2
  Alopecia | 4
  Anal Hemorrhage | 1
  Anemia | 6
  Anorexia | 20
  Anxiety | 2
  Arthralgia | 12
  Arthritis | 2
  Back Pain | 9
  Bacteremia | 1
  Belching | 1
  Blepharitis | 1
  Bloating | 3
  Blurred Vision | 14
  Body Aches | 1
  Bone Pain | 2
  Burning Eyes | 1
  Callus Tenderness | 1
  Cataract | 6
  Cheilitis | 1
  Cholesterol High | 1
  Choroid Mild Tortuosity | 1
  Chronic Kidney Disease | 4
  Constant Eye Pressure | 1
  Constipation | 21
  Corneal Abrasion | 4
  Corneal Ulcer | 1
  Corners of Mouth Cracking Open | 1
  Cotton Wool Spot | 1
  Cough | 3
  Covid-19 | 2
  Crawling Sensation on Skin | 1
  Creatinine Increased | 2
  Dehydration | 5
  Depression | 10
  Dermatochalasis | 1
  Diarrhea | 14
  Diplopia | 1
  Dizziness | 2
  Dry Eye | 12
  Dry Mouth | 11
  Dry Nose | 1
  Dry Skin | 6
  Dry Throat | 1
  Dysgeusia | 16
  Dyspnea | 16
  Dysuria | 1
  Ear Pain | 1
  Edema Face | 2
  Edema Limbs | 9
  Edema Trunk | 2
  Epigastric Discomfort | 1
  Epistaxis | 5
  Eye Infection | 1
  Eye Redness | 2
  Eyelash Epilation | 1
  Fall | 10
  Fatigue | 56
  Fever | 3
  Flank Pain | 5
  Flatulence | 1
  Floaters | 3
  Flu Like Symptoms | 1
  Fracture | 1
  Gait Disturbance | 3
  Gastroenteritis | 1
  Gastritis | 1
  Gastroesophageal Reflux Disease | 7
  Gastrointestinal Pain | 1
  Gastrointestinal Reflux Disease | 1
  Generalized Weakness | 1
  Glaucoma | 1
  Gritty Eyes | 1
  Headache | 6
  Hematuria | 1
  Hemorrhoidal Hemorrhage | 2
  Hoarseness | 1
  Hypercalcemia | 4
  Hyperglycemia | 5
  Hyperphosphatemia | 8
  Hypertension | 2
  Hypertrichosis | 1
  Hypertriglyceridemia | 8
  Hypoalbuminemia | 5
  Hypocalcemia | 1
  Hyponatremia | 7
  Hypophosphatemia | 5
  Hypotension | 4
  Hypothyroidism | 1
  Hypoxemia Post Monoclonal Antibody Infusion | 1
  Insomnia | 6
  Intermittent Phlegm | 1
  Keratitis | 6
  Keratopathy | 1
  Lip Blister | 1
  Lipase Increased | 2
  Localized Edema | 3
  Lymphocyte Count Decreased | 1
  Melena | 2
  Memory Impairment | 1
  Metavirus | 1
  Mucositis oral | 26
  Muscle Aches | 1
  Muscle Cramp | 13
  Myalgia | 2
  Nail Changes | 11
  Nail Discoloration | 5
  Nail Lifting | 9
  Nail Loss | 10
  Nail Ridges | 4
  Nasal Congestion | 3
  Nasal Mucosa Irritation | 1
  Nasal Sores | 1
  Nausea | 19
  Neck Pain | 2
  Non-cardiac Chest Pain | 2
  Non-neurovascular Age Related Macular Degeneration | 1
  Onychauxis | 1
  Oral Dysesthesia | 1
  Oral Pain | 2
  Otitis Externa | 1
  Overactive Bladder | 1
  Pain in Extremity | 19
  Pain of Skin | 3
  Pain | 28
  Palmar-plantar Erythrodysesthesia Syndrome | 6
  Paresthesia | 1
  Paronychia | 9
  Pelvic pain | 1
  Periorbital Edema | 1
  Peripheral Motor Neuropathy | 2
  Peripheral Sensory Neuropathy | 21
  Platelet Count Decreased | 2
  Pleural effusion | 3
  Pneumonia | 1
  Port Site Redness | 1
  Posterior Vitreous Detachment Posterior Vitreous Detachment | 1
  Presbyopia | 1
  Productive Cough | 5
  Pruritus | 1
  Pseudophakia | 2
  Punctate Keratopathy | 1
  Rash Maculo-papular | 6
  Rash | 2
  Rectovaginal Fistula | 1
  Retinal Hemorrhage | 1
  Retinal Vascular Disorder | 1
  Retinopathy | 2
  Rhinitis Sicca | 1
  Shingles | 1
  Sinus Tachycardia | 2
  Small Intestinal Obstruction | 2
  Sore Throat | 6
  Syncope | 1
  Teeth Extraction | 1
  Thromboembolic Event | 1
  Thrush | 2
  Toe Intermittent Drainage | 1
  Tooth Infection | 1
  Tremor | 1
  Trichiasis | 2
  Trichomegaly | 1
  Trochanteric Bursitis | 1
  Vaginal Discharge | 1
  Vaginal Pain | 2
  Vomiting | 12
  Watering Eyes | 8
  Weight Gain | 4
  Weight Loss | 23
  Wheezing | 1

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Treatment (Infigratinib)
All-Cause Mortality (participants affected / at risk) | 13/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Infigratinib) (N=17)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Covid-19 (Immune system disorders) | 1 (1)
Gasteroenteritis (Gastrointestinal disorders) | 1 (1)
Metavirus (Infections and infestations) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Infigratinib) (N=17)
Teeth Extraction (Gastrointestinal disorders) | 1 (1)
Abdominal Cramping (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 9 (18)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 2 (3)
Allergic Reaction (Immune system disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Anorexia (Metabolism and nutrition disorders) | 11 (20)
Anxiety (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (12)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Bacteremia (Infections and infestations) | 1 (1)
Belching (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Hypoxemia Post Monoclonal Antibody Infusion (Blood and lymphatic system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 8 (14)
Body Aches (General disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cataract (Eye disorders) | 4 (6)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Cholesterol High (Investigations) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 2 (4)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 13 (21)
Corneal Ulcer (Eye disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Creatinine Increased (Investigations) | 2 (2)
Platelet Count Decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Depression (Psychiatric disorders) | 8 (10)
Diarrhea (Gastrointestinal disorders) | 9 (14)
Dizziness (Nervous system disorders) | 2 (2)
Dry Eye (Eye disorders) | 8 (12)
Dry Mouth (Gastrointestinal disorders) | 10 (11)
Dry Skin (Skin and subcutaneous tissue disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 9 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (16)
Dysuria (Renal and urinary disorders) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 1 (1)
Edema Limbs (General disorders) | 5 (9)
Edema Trunk (General disorders) | 2 (2)
Edema Face (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Eye Redness (Eye disorders) | 2 (2)
Burning Eyes (Eye disorders) | 1 (1)
Choroid Mild Tortuosity (Eye disorders) | 1 (1)
Trichiasis (Eye disorders) | 2 (2)
Corneal Abrasion (Eye disorders) | 1 (4)
Cotton Wool Spot (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Punctate Keratopathy (Eye disorders) | 1 (1)
Gritty Eyes (Eye disorders) | 1 (1)
Posterior Vitreous Detachment (Eye disorders) | 1 (1)
Retinal Hemorrhage (Eye disorders) | 1 (1)
Trichomegaly (Eye disorders) | 1 (1)
Blepharitis (Eye disorders) | 1 (1)
Constant Eye Pressure (Eye disorders) | 1 (1)
Pseudophakia (Eye disorders) | 1 (2)
Presbyopia (Eye disorders) | 1 (1)
Dermatochalasis (Eye disorders) | 1 (1)
Keratopathy (Eye disorders) | 1 (1)
Eye Infection (Eye disorders) | 1 (1)
Eyelash Epilation (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (10)
Fatigue (General disorders) | 17 (56)
Fever (General disorders) | 2 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Flatulence (Gastrointestinal disorders) | 1 (1)
Floaters (Eye disorders) | 3 (3)
Flu Like Symptoms (General disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gait Distrubance (General disorders) | 1 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 6 (7)
Dry Nose (Gastrointestinal disorders) | 1 (1)
Rectovaginal Fistula (Gastrointestinal disorders) | 1 (1)
Dry Throat (Gastrointestinal disorders) | 1 (1)
Epigastric Discomfort (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Reflux Disease (Gastrointestinal disorders) | 1 (1)
Generalized Weakness (General disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (6)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Anal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (5)
Hyperphosphatemia (Metabolism and nutrition disorders) | 7 (8)
Hypertension (Vascular disorders) | 2 (2)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (5)
Hypotension (Vascular disorders) | 3 (4)
Hypothyroidism (Endocrine disorders) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (6)
Intermittent Phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Keratitis (Eye disorders) | 2 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Lipase Increased (Investigations) | 2 (2)
Localized Edema (General disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (1)
Melena (Gastrointestinal disorders) | 2 (2)
Memory Impairment (Nervous system disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (26)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 5 (13)
Muscle Aches (Musculoskeletal and connective tissue disorders) | 1 (1)
Trochanteric Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nail Changes (Skin and subcutaneous tissue disorders) | 9 (11)
Nail Discoloration (Skin and subcutaneous tissue disorders) | 5 (5)
Nail Lifting (Skin and subcutaneous tissue disorders) | 5 (9)
Nail Loss (Skin and subcutaneous tissue disorders) | 3 (10)
Nail Ridges (Skin and subcutaneous tissue disorders) | 4 (4)
Nasal Sores (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (19)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Non-cardiac Chest Pain (General disorders) | 2 (2)
Non-neurovascular Age Related Macular Degeneration (Eye disorders) | 1 (1)
Onychauxis (Skin and subcutaneous tissue disorders) | 1 (1)
Oral Dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 2 (2)
Otitis Externa (Infections and infestations) | 1 (1)
Overactive Bladder (Renal and urinary disorders) | 1 (1)
Pain of Skin (Skin and subcutaneous tissue disorders) | 3 (3)
Pain (General disorders) | 8 (28)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 (19)
Palmar-plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 3 (6)
Paresthesia (Nervous system disorders) | 1 (1)
Paronychia (Infections and infestations) | 5 (9)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 14 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Port Site Redness (General disorders) | 1 (1)
Rhinitis Sicca (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retinal Vascular Disorder (Eye disorders) | 1 (1)
Retinopathy (Eye disorders) | 2 (2)
Shingles (Infections and infestations) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 2 (2)
Lip Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Crawling Sensation on Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Callus Tenderness (Skin and subcutaneous tissue disorders) | 1 (1)
Corners of Mouth Cracking Open (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal Mucosa Irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Toe Intermittent Drainage (Skin and subcutaneous tissue disorders) | 1 (1)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
Thrush (Infections and infestations) | 2 (2)
Tooth Infection (Infections and infestations) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (12)
Watering Eyes (Eye disorders) | 8 (8)
Weight Gain (Investigations) | 1 (4)
Weight Loss (Investigations) | 11 (23)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT04233567/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04233567/ICF_000.pdf